CLINICAL TRIAL: NCT01788631
Title: A Phase II, Randomized, Placebo-Controlled Trial of Regadenoson in Sickle Cell Anemia
Brief Title: A Phase II Trial of Regadenoson in Sickle Cell Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); La Jolla Institute for Allergy & Immunology (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Washington University School of Medicine (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Illinois at Chicago (Other); Medical College of Wisconsin (Other); Duke University (Other); Johns Hopkins University (Other); Wayne State University (Other); Baylor College of Medicine (Other); UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Principal Investigator, David G. Nathan, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-005; 1P50HL110790-01 (NIH)
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — regadenoson; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regadenoson Arm (Active Comparator): 1.44 mcg/kg/hour infused over 48 hours
  Interventions: Drug: Regadenoson
- Placebo Arm (Placebo Comparator): Placebo infused over 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regadenoson — Regadenoson is an A2AR agonist that is a coronary vasodilator. It is chemically described as adenosine, 2-[4-[(methylamino)carbonyl]-1H-pyrazol-1-yl]-, monohydrate. Its molecular formula is C15H18N8O5. Regadenoson has an FDA indication for use in radionuclide myocardial perfusion imaging in patients unable to undergo adequate exercise stress. It has lower affinity for non-A2A adenosine receptor subtypes thought to be associated with some of the adverse effects associated with non-selective adenosine receptor agonists, which increase extracellular adenosine by blocking its uptake into cells. The maximal plasma concentration of regadenoson is achieved within 1 to 4 minutes after injection and parallels the onset of the pharmacodynamic response. Its half-life is approximately 2 to 4 minutes.
  Other Names: Lexiscan
  Arms: Regadenoson Arm
Drug: Placebo — This study uses 0.9% Normal Saline (NS) as placebo. This is a sterile sodium chloride solution usually used to replenish fluids and electrolytes. It contains no additives, and is a standard solution used as placebo in clinical trials where the study drug is administration intravenously. NS will be prepared by investigational pharmacy.
  Other Names: Regadenoson Placebo, Lexiscan Placebo, 0.9% Normal Saline
  Arms: Placebo Arm

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug called Regadenoson (or Lexiscan) to learn whether the drug works in treating a specific disease, in this case Sickle Cell Disease (SCD). "Investigational" means that the drug is being studied. It also means that the FDA has not yet approved the drug for your type of disease.

SCD is an inherited blood disorder that causes the red blood cells to change their shape from a round shape to a half-moon/crescent or sickled shape. People who have SCD have a different type of protein that carries oxygen in their blood (hemoglobin) than people without SCD. This different type of hemoglobin makes the red blood cells change into crescent shape under certain conditions. Sickle-shaped cells are a problem because they often get stuck in the blood vessels blocking the flow of blood, and cause inflammation and injury to important areas in the body.

Regadenoson (trade name Lexiscan) is a drug that may prevent this inflammation and injury caused by the sickle shaped cells. This drug is approved by the FDA to be used as a fast infusion during a heart stress test in people who are unable to exercise enough to put stress on their heart by making the heart beat faster. Regadenoson has been studied as a long infusion at this dose in adults, and no safety issues have been identified (ClinicalTrials.gov Identifier: NCT01085201). This is the first study to look at patient benefit with the long infusion of the drug. This drug has been used in laboratory experiments and information from those other research studies suggests that this drug may help to protect the body from damage caused by sickle-shaped cells in this research study.

In this research study, the investigators are specifically looking to see if Regadenoson is an effective treatment for pain crises and acute chest syndrome in SCD.

DETAILED DESCRIPTION:
If you are willing to participate in this research study you will be asked to undergo some screening tests and procedures to confirm your eligibility. Many of these tests and procedures are likely to be part of regular sickle cell anemia care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests and procedures recently, they may or may not have to be repeated. The tests and procedures include: a medical history, physical examination, blood tests, blood or urine pregnancy test (if applicable) and an electrocardiogram. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in the research study. At the time of screening we will also ask you about your pain level.

Because no one knows which of the study options is best, you will be "randomized" into one of the study groups: the "study drug" group, which will receive Regadenoson, or the "control" group, which will receive placebo. Randomization means that you are put into a group by chance. It is like flipping a coin. Neither you nor the research doctor will choose what group you will be in. You will have an equal (50/50) chance of being placed in either group. Neither you nor the research doctor will know what group you are in.

You will be given a study medication and it will contain either Regadenoson or placebo (fluids with no medicine).

You will be given one infusion of the study drug while you are admitted to the hospital for a pain crisis. The study drug will be infused with fluids. You will stay in the hospital for at least 3 days and 2 nights. Your infusion will be 48 hours long, followed by a 6-hour observation period. During your infusion, you will receive standard treatment for your pain crisis. The study drug will be given through a separate part of your body from the infusions that are part of your standard treatment. The study drug will not be available after your participation in the study ends.

Before the infusion: We will place a small tube in your vein called an IV, which will be used only to infuse the study drug. It will not be used for infusions that are part of standard treatment for your pain crisis. During the study drug infusion, standard treatment will be given through a separate IV. We can use your standard treatment IV or a needle to draw blood for the required blood test. If it is hard to draw blood from your veins, we may ask you if you would like to use a peripherally inserted central catheter (PICC line) for your blood draws. A PICC line is a small tube that is placed in a vein in your arm and goes through to a vein in your chest. A chest x-ray is usually done to make sure it is in the right veins. It is your choice to decide whether you would like to use a PICC line. We will record your blood pressure and heart rate every 5-10 minutes, until they have stabilized. We will also ask you about your pain level at the time of your blood test.

During the 48 hour infusion: Your heart rate and the amount of oxygen in your blood will be monitored continuously using a device that fits over your finger. We will take about 2-3 teaspoons of blood at 24 and 48 hours after the beginning of your infusion for tests to try to understand how the drug affects your body. We will ask you about your pain level at the time of each blood test. We will take your blood pressure every 30 minutes for the first 2 hours, then every hour for the next two hours, then every 2 hours for the remainder of the infusion.

A six hour observation period will take place immediately after the infusion. At this time you will undergo the following: your heart rate and the amount of oxygen in your blood will be monitored continuously with a device that fits over your finger. We will take about 5 teaspoons of blood at the end of the period to try to understand how the study drug affects your body. We will ask you about your pain level at the time of your blood test. We will take your blood pressure every 2 hours for the full duration of the observation period.

You may not eat or drink anything that contains caffeine, such as coffee, tea, chocolate or sodas during the infusion and observation periods.

We would like to keep track of your medical condition for 30 days after you receive the study drug. We would like to do this by contacting you on the telephone weekly during the 30 days after your participation to see how you are doing.

ELIGIBILITY:
Inclusion Criteria:

* Must have sickle cell anemia confirmed by hemoglobin analysis
* Must be admitted to hospital for pain or ACS
* Reliable IV access as determined by the study physician
* Participants must have the laboratory indices as defined below:

  * Hemoglobin ≥ 5 g/dL
  * Platelets > 100,000/mcL
  * ALT (SGPT) < 3 X institutional upper limit of normal
  * Serum creatinine ≤ 1.5 mg/dL
  * INR ≤2.0, PTT ≤ 48 seconds

Exclusion Criteria:

* Pregnant or breastfeeding
* Current physician diagnosis of asthma defined by treatment with systemic corticosteroids within the last 12 months or predicted/current use of asthma controller medications
* 10 or more hospitalizations for pain in the last 12 months
* Receiving regularly scheduled transfusions
* Severe ACS
* Second or third degree AV block or sinus node dysfunction
* History of a bleeding diathesis
* History of clinically overt stroke within 3 years
* History of severe hypertension not adequately controlled with anti-hypertensive medications
* Receiving chronic anti-coagulation or anti-platelet therapy
* History of metastatic cancer
* Receiving any other study agents or have received a study agent in the past 30 days
* Uncontrolled intercurrent illness
* Known HIV
* Have previously enrolled and received the investigational agent as part of this study
* Taking medications that may interact with the investigational agent
* Have previously undergone a hematopoietic stem cell transplant or solid organ transplant

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11-10 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Nathan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Field JJ, Majerus E, Gordeuk VR, Gowhari M, Hoppe C, Heeney MM, Achebe M, George A, Chu H, Sheehan B, Puligandla M, Neuberg D, Lin G, Linden J, Nathan DG. Randomized phase 2 trial of regadenoson for treatment of acute vaso-occlusive crises in sickle cell disease. Blood Adv. 2017 Aug 28;1(20):1645-1649. doi: 10.1182/bloodadvances.2017009613. eCollection 2017 Sep 12. PMID 29296811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2013 and November 2016, 4,940 hospital admissions were screened to enroll 100 study subjects. Patients were recruited at the time of sickle cell vaso-occlusive crises in outpatient clinics, emergency departments, and inpatient units.
Pre-assignment Details: Prior to study arm randomization and assignment, patients were screened using the following testing methods: Confirmation of sickle cell genotype, complete blood count with differential, chemistry, coagulation testing (Including PTT, and INR), and pregnancy testing for female participants.
Period: Overall Study
Arm/Group | Regadenoson Arm | Placebo Arm
Started | 52 | 44
Randomized | 53 | 47
Completed | 49 | 43
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regadenoson Arm | Placebo Arm | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Continuous [Median (Full Range); unit: years] | 25 [10 to 54] | 26 [13 to 56] | 25 [10 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 31 | 23 | 54
Region of Enrollment [Number; unit: Participants]
  United States | 53 | 47 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Invariant Natural-Killer T-Cell (iNKT Cell) Activation by 70% or More
Description: To determine if infusional Regadenoson reduced iNKT cell activation among individuals with sickle cell anemia (SCA) and pain or acute chest syndrome (ACS) compared to placebo by 70% or greater.
Time Frame: Baseline-End of study infusion over 48 hours
Population: Treated patients with baseline and end of infusion blood samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
Participants | 21 | 10

2. Secondary Outcome: Length of Hospital Stay
Description: To determine if regadenoson reduces length of hospital stay among individuals admitted with SCA and pain or ACS compared to placebo
Time Frame: Hospital Presentation- Hospital Discharge, assessed up to 1 month
Population: All patients who had baseline and end of infusion blood samples.
Measure: Median (Full Range); unit: Days
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
Days | 3.96 [2.23 to 19.25] | 3.99 [2.34 to 30.40]

3. Secondary Outcome: Number of Participants With an Improvement in Respiratory Symptoms
Description: To determine if regadenoson improved respiratory symptoms among individuals with sickle cell anemia (SCA) and pain or acute chest syndrome (ACS) compared to placebo. Patients were classified as having an improvement in respiratory symptoms if they experienced any of the following outcomes:(1) respiratory rate decreased by 25% from baseline or normalized (≤20 bpm) or (2) degree of hypoxia (SpO2) on room air increased by 10% from baseline or normalized (≥92%) or (3) thoracic pain improved by 3 points from baseline on a 10-point visual analog scale.
Time Frame: Baseline-End of study infusion over 48 hours
Population: All patients who had baseline and end of infusion blood samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
Participants | 10 | 9

4. Secondary Outcome: Opioid Use
Description: To determine if regadenoson reduces opioid use among individuals with SCA and pain or ACS compared to placebo.
Time Frame: Baseline-End of study infusion over 48 hours
Population: All patients who had baseline and end of infusion blood samples.
Measure: Median (Full Range); unit: mg/kg/hr
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
mg/kg/hr | 0.03 [0.00 to 0.50] | 0.04 [0.00 to 0.36]

5. Secondary Outcome: Level of Inflammatory Markers (A2A)
Description: To determine if regadenoson reduces levels of inflammatory markers among individuals with SCA and pain or ACS compared to placebo.
Time Frame: Baseline-End of study infusion over 48 hours
Population: All patients who had baseline and end of infusion blood samples.
Measure: Median (Full Range); unit: A2A levels as percent of baseline
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
A2A levels as percent of baseline | 86.39 [35.3 to 316.67] | 100.95 [17.44 to 404.66]

6. Secondary Outcome: Level of Inflammatory Markers (IL-4)
Description: as for outcome 5
Time Frame: Baseline-End of study infusion over 48 hours
Population: All patients who had baseline and end of infusion blood samples.
Measure: Median (Full Range); unit: IL-4 levels as percent of baseline
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
IL-4 levels as percent of baseline | 85.89 [33.51 to 389.76] | 100.91 [17.35 to 351.09]

7. Secondary Outcome: Level of Inflammatory Markers (IFN-gamma)
Description: as for outcome 5
Time Frame: Baseline-End of study infusion over 48 hours
Population: All patients who had baseline and end of treatment samples
Measure: Median (Full Range); unit: IFN-gamma levels as percent of baseline
Arm/Group | Regadenoson Arm | Placebo Arm
Number analyzed (Participants) | 49 | 43
IFN-gamma levels as percent of baseline | 97.38 [42.50 to 293.83] | 105.66 [28.01 to 420.99]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time patients presented to the emergency department for their vaso-occlusive crisis through 30 days post- hospital discharge.
Description: For this study, all adverse events Grade 3 and above were categorized as serious adverse events.
Arm/Group | Regadenoson Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/44
Serious Adverse Events (participants affected / at risk) | 14/52 | 16/44
Other Adverse Events (participants affected / at risk) | 44/52 | 35/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regadenoson Arm (N=52) | Placebo Arm (N=44)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Blood bilirubin increased (Investigations) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Hemoglobin increased (Investigations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Pain (General disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regadenoson Arm (N=52) | Placebo Arm (N=44)
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 4 | 5
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 | 0
Blurred vision (Eye disorders) | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Chills (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Delirium (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 0
Dry eye (Eye disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Fever (General disorders) | 7 | 6
Flushing (Vascular disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 10
Hematuria (Renal and urinary disorders) | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Ileus (Gastrointestinal disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2
Infusion related reaction (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Lethargy (Nervous system disorders) | 2 | 0
Localized edema (General disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 5 | 11
Non-cardiac chest pain (General disorders) | 0 | 4
Pain (General disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 7
Palpitations (Cardiac disorders) | 0 | 2
Photophobia (Eye disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Scleral disorder (Eye disorders) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No